CLINICAL TRIAL: NCT03096041
Title: Phase 3 Study Randomized Against Placebo, Evaluating the Efficacy of Auriculotherapy in Patients With Musculoskeletal Pain by Aromatase Inhibitors in Adjuvant Treatment of Breast Cancer (TRIPLE-A)
Brief Title: Phase 3 Study Randomized Evaluating the Efficacy of Auriculotherapy in Patients With Musculoskeletal Pain by Aromatase Inhibitors
Acronym: TRIPLE-A
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Francois Baclesse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: TRIPLE-A
Record Dates: First submitted 2017-03-20; First posted 2017-03-30 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Musculoskeletal Pain; Breast Cancer
Keywords: auriculotherapy; aromatase inhibitors; adjuvant treatment
MeSH Terms: conditions — Musculoskeletal Pain; Breast Neoplasms | interventions — Auriculotherapy

STUDY DESIGN:
Who Masked: Participant
Masking Description: Single blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental arm (Experimental): Auriculotherapy for analgesic use
  Interventions: Device: Auriculotherapy for analgesic use
- Controle arm (Placebo Comparator): Placebo auriculotherapy
  Interventions: Device: Placebo auriculotherapy

INTERVENTIONS:
Device: Auriculotherapy for analgesic use — The ASP will be applied to specific pain points
  Arms: Experimental arm
Device: Placebo auriculotherapy — The ASP will be applied to placebo points (not specific to pain)
  Arms: Controle arm

SUMMARY:
Auriculotherapy is a complementary medicine, with few side effects, without contraindication, inexpensive and not very restrictive.Its efficacy has been found in several tests especially for the treatment of intraoperative pain. It remains more controversial in other indications. Evaluation of the value of auriculotherapy is often difficult because of the methodological limitations of the trials conducted. In the daily practice, the auriculotherapy is proposed to improve the articular pains of patients treated by AA. This Phase III study aims at validate this approach.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years of age
* Patients with anti-aromatases in adjuvant treatment of breast cancer
* Menopausal women
* Treatment with aromatase inhibitors (anti-aromatase, AA) initiated for more than 3 months. In the case of a change in anti-aromatase, the last treatment must be started for more than 3 months.
* Musculoskeletal pain appearing or increased under AA:
* Overall pain score of QCD ≥3 (on a scale of 0 to 10)
* Pain on at least 2 sites
* Pain for at least 3 months
* History of radiotherapy and / or adjuvant chemotherapy authorized
* Patients may have received tamoxifen
* Patient affiliated to a social security system
* Patient mastering the French language and able to complete the evaluation questionnaires
* Free and Informed Consent

Exclusion Criteria:

* Patients who have already undergone treatment in auriculotherapy for the same indication
* Patient benefiting at the same time from a PNCAVT (acupuncture or homeopathy) for musculoskeletal pain
* Wearing hearing aids hindering the placement of semi-permanent needles (ASP)
* Wearing of a valve prosthesis
* Patient under guardianship or unable to give informed consent
* Patient unable to undergo medical follow-up for geographical, social or psychopathological reasons

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 197 (Actual)
Dates: Start 2017-07-05 (Actual); Primary Completion 2025-07-07 (Actual); Study Completion 2025-07-07 (Actual)

PRIMARY OUTCOMES:
Decrease in the overall pain score | 3 months after auriculotherapy initiation
  The proportion of patients with a 2-point or greater decrease in the overall pain

CONTACTS AND LOCATIONS:
Locations (7):
- France (7):
  - Centre François Baclesse, Caen
  - Hôpital Privé Paul d'Egine, Champigny-sur-Marne
  - Hôpital Cognac-Jay - Forcilles, Férolles-Attilly
  - CHU Grenoble, Grenoble
  - Centre Oscar Lambret, Lille
  - Groupe Hospitalier Paris St Joseph, Paris
  - IGR, Villejuif

IPD SHARING:
Plan to Share IPD: No